CLINICAL TRIAL: NCT06841653
Title: A.I and Machine Learning Based Risk Prediction Model to Improve the Clinical Management of Endometrial Cancer: a Composite Approach Integrating the MultiOMics IMmune-IConographic Pattern (MOMIMIC Score) Towards Precision Oncology and Surgery.
Brief Title: A.I and Machine Learning Based Risk Prediction Model to Improve the Clinical Management of Endometrial Cancer.
Status: Recruiting | Type: Observational
Sponsor: Regina Elena Cancer Institute (Other)
Collaborators: University of Rome Tor Vergata (Other); Casa Sollievo della Sofferenza-IRCCS, San Giovanni Rotondo (Unknown); Universita degli Studi di Palermo (Other)
Responsible Party: Sponsor
Other Study IDs: RS203/IRE/24
Record Dates: First submitted 2025-02-18; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Endometrium Cancer
Keywords: MultiOMics IMmune-IConographic pattern
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Tissue samples and peripheral venous blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective cohort: Fresh tissue samples stored at -80°C, collected at the Institute's IRE Biobank (a starting from 2019) and tissue preserved in paraffin at the biobank at 4°C at the UOC Pathological Anatomy archive, for carrying out WES, RNA-seq, scRNA-seq, spatial transcriptomics, metabolomics, proteomics, digital pathology, immune infiltrate characterization (e.g. FACS, immunohistochemistry)
- Prospective cohort: Collection of tissue samples obtained at the time of surgery and verified by the anatomical pathologist for the actual availability and adequacy, for the purpose of the creation of organoids (Patient-Derived Organoids, PDO), cell lines and co-cultures (created with the patient's own peripheral immune cells, collected and processed), in the context of which secretomics analyzes will be conducted using Olink and Luminex.

SUMMARY:
Prediction of preoperative endometrial biopsy: the evolution from hyperplasia to cancer, the prognosis and the risk of recurrence. Intelligence methods artificial risk will be used to redefine the current risk classes including our profile immuno-mutational to provide a more precise characterization and closer to the real prognosis of the patient.

DETAILED DESCRIPTION:
Identify new risk factors for endometrial cancer, using an integrated multi-omics approach linked to a specific immune pattern (called MOMIMIC score) useful for improving oncology and surgery precision. The aim is to evaluate the predictive value of the MOMIMIC score for early identification of progression from precancerous lesions to endometrial carcinoma, prognosis and relapses, to help the clinician in the decision to treatments. Through the identification during hysteroscopy of the most appropriate site for biopsies targeted endometrials, through an artificial intelligence algorithm applied to the video system hysteroscopic which, by comparing the information from the omics approach and the hysteroscopic image combined with radiogenomic information, it could help the gynecologist in the procedure and provide information on the prognosis through the omics-iconographic profile in order to calculate a preoperative predictive score. Furthermore by modulating the surgical radicality, according to the information obtained, there will be a tendency to preserve fertility in young patients with a low-risk profile (since currently the risk factors are not sufficient to discriminate for a non-treatment radical). This will help the surgeon through an artificial intelligence algorithm applied to the system robotic/laparoscopic video, will guide the operator in decision-making procedures regarding the resection margins tumor, metastasis localization, pathological lymph node detection, and imaging driven by biomolecular information.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years;
* Histological diagnosis of endometrial hyperplasia, endometrioid adenocarcinoma of the endometrium, healthy endometrium in patients undergoing total hysterectomy for benign extra-endometrial disease;
* Written informed consent (to the study and data processing), for the party's patients only prospective and/or in follow-up) For the retrospective cohort: availability of samples adequately stored at the biobank of the Institute and availability of data relating to follow-up (at least 2 years)

Exclusion Criteria:

All exclusion criteria adopted in the surgical protocols will be applied to the study. In particular:

* Comorbidities not controlled with adequate medical therapy;
* Infections of the endometrial cavity (pyometra);
* Synchronous cancer;
* Neoadjuvant treatments;
* Previous radiotherapy treatments of the pelvic region;
* Hormone therapies.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — * patients undergoing hysterectomy for benign extra-endometrial pathology;
  * patients diagnosed with endometrial hyperplasia without atypia;
  * patients diagnosed with endometrial hyperplasia without atypia;
  * patients diagnosed with endometrial carcinoma of the endometrioid histology at any stage disease;
Study Population: Patients suffering from endometrial cancer.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2026-06-20 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
OS (overall survival) | 24 months
  The study will evaluate the predictive value of the MultiOMics-IMmune-Iconographic model (global mutational profiling, RNA-seq of single cells coupled with the Spatial transcriptomics, proteomic and metabolomic profile) following the data obtained from the identification of new risk factors for endometrial carcinoma, in patients at high or low risk. They will be tested from Random Survival Forest to determine how capable a feature is discriminate between the 4 groups in terms of OS (overall survival). The selected features will be used in combination with the known prognostic clinical and histopathological risk factors described by ESMO-ESGO-ESTRO.
DSF (disease-free survival) | 24 months
  The study will evaluate the predictive value of the MultiOMics-IMmune-Iconographic model (global mutational profiling, RNA-seq of single cells coupled with the Spatial transcriptomics, proteomic and metabolomic profile) following the data obtained from the identification of new risk factors for endometrial carcinoma, in patients at high or low risk.
  They will be tested via Random Survival Forest to determine how capable a feature is discriminate between the 4 groups in terms of impact on progression to cancer, recurrence, DFS (disease-free survival).

SECONDARY OUTCOMES:
Area under the curve (AUC) | 24 months
  In order to obtain a more robust estimate of accuracy of the MultiOMics-IMmune predictive signature, for validation, we will use two groups of patients composed of a minimum of 200 cases (100 high risk and 100 low risk), at a reduction from 30% confidence interval to 95% when signature performance are kept constant. Considering the area under the curve (AUC).
Accuracy (ACC) | 24 months
  In order to obtain a more robust estimate of accuracy of the MultiOMics-IMmune predictive signature, for validation, we will use two groups of patients composed of a minimum of 200 cases (100 high risk and 100 low risk), at a reduction from 30% confidence interval to 95% when signature performance are kept constant. Considering Accuracy (ACC).

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS National Cancer Institute "Regina Elena", Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided